CLINICAL TRIAL: NCT03433274
Title: Clinical Trial to Evaluate the Safety and Effectiveness of Using the Tendyne Transcatheter Mitral Valve System for the Treatment of Symptomatic Mitral Regurgitation
Acronym: SUMMIT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CS0004-P
Record Dates: First submitted 2018-02-08; First posted 2018-02-14 (Actual); Results first posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Mitral Regurgitation; Mitral Insufficiency; Mitral Valve Insufficiency; Cardiovascular Diseases; Valve Disease, Heart; Heart Valve Diseases; Functional Mitral Regurgitation; Degenerative Mitral Valve Disease
MeSH Terms: conditions — Mitral Valve Insufficiency; Cardiovascular Diseases; Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (5):
- Randomized Cohort - Treatment Group (Experimental): Treatment of mitral regurgitation with the Tendyne Transcatheter Mitral Valve System
  Interventions: Device: Tendyne Mitral Valve System
- Randomized Cohort - Control Group (Active Comparator): Treatment of mitral regurgitation within commercially approved MitraClip system indications
  Interventions: Device: MitraClip System
- Non-repairable Cohort (Experimental): Treatment of mitral regurgitation with the Tendyne Transcatheter Mitral Valve System
  Interventions: Device: Tendyne Mitral Valve System
- Severe Mitral Annular Calcification (MAC) Cohort (Experimental): Treatment of mitral regurgitation and mitral annular calcification with the Tendyne Transcatheter Mitral Valve System
  Interventions: Device: Tendyne Mitral Valve System
- Severe Mitral Annular Calcification Continued Access Plan (MAC CAP) Cohort (Experimental): Treatment of mitral regurgitation and mitral annular calcification with the Tendyne Transcatheter Mitral Valve System after the completion of enrollment in the Severe MAC Cohort
  Interventions: Device: Tendyne Mitral Valve System

INTERVENTIONS:
Device: Tendyne Mitral Valve System — Mitral valve replacement
  Arms: Non-repairable Cohort; Randomized Cohort - Treatment Group; Severe Mitral Annular Calcification (MAC) Cohort; Severe Mitral Annular Calcification Continued Access Plan (MAC CAP) Cohort
Device: MitraClip System — Percutaneous mitral valve repair using the MitraClip system.
  Arms: Randomized Cohort - Control Group

SUMMARY:
Prospective, controlled, multicenter clinical investigation with four trial cohorts: Randomized, Non-repairable, Severe Mitral Annular Calcification (MAC) and Severe Mitral Annular Calcification Continued Access Plan (MAC CAP). Subjects in the Randomized cohort were randomized in a 1:1 ratio to the trial device or to the MitraClip system. Subjects in the Non-repairable, Severe MAC, and Severe MAC CAP cohorts were receive the trial device.

The objective of the Clinical Trial to Evaluate the Safety and Effectiveness of Using the Tendyne Transcatheter Mitral Valve System for the Treatment of Symptomatic Mitral Regurgitation (SUMMIT) was to evaluate the safety and effectiveness of the Tendyne Transcatheter Mitral Valve System for the treatment of patients with symptomatic, moderate-to-severe or severe mitral regurgitation or for patients with symptomatic mitral valve disease due to severe mitral annular calcification.

This randomized controlled trial would provide the opportunity to evaluate the safety and clinical benefits of the Tendyne Transcatheter Mitral Valve System compared to the MitraClip System in patients with symptomatic, moderate-to-severe or severe mitral regurgitation, within approved MitraClip indications. In addition, the safety and effectiveness of the Tendyne Transcatheter Mitral Valve System would be evaluated in patients with severe mitral annular calcification who are at prohibitive risk for mitral valve surgery. Patients who were not suitable for mitral valve surgery for reasons other than severe mitral annular calcification and were also not suitable for transcatheter repair with MitraClip, would be enrolled in the Non-repairable cohort.

Subjects would be seen at screening, pre- and post-procedure, discharge, 30 days, 3 months, 6 months, and annually through 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic, moderate-to-severe or severe mitral regurgitation (MR ≥ Grade III per American Society of Echocardiography criteria), or severe mitral annular calcification (MAC), where a transcatheter therapy is deemed more appropriate than open surgery by the local site heart team.

   Note: MR and MS severity must be determined by assessment of a qualifying transesophageal echocardiogram (TEE) and transthoracic echocardiogram (TTE), obtained within 120 days prior to subject consent, and must be confirmed by the Echocardiography Core Laboratory.

   Note: Patients with severe MAC must have symptomatic mitral valve disease associated with MR≥ Grade III, or severe mitral stenosis (MS), or both moderate MR and moderate MS as assessed by the Echocardiography Core Laboratory.
2. NYHA Functional Classification ≥ II (if Class IV, patient must be ambulatory).
3. The local site heart team determines that the subject has been adequately treated per applicable standards for coronary artery disease (e.g., revascularization), left ventricular dysfunction (e.g., cardiac resynchronization therapy) and heart failure (e.g., GDMT). The SEC must concur that the subject has been adequately treated.
4. The local site heart team and the SEC concur on the intended study cohort for the subject.

   Randomized cohort: Eligibility for this cohort is limited to subjects where the local site heart team deems the mitral valve anatomy is suitable for TEER and are within approved Mitra Clip indications, which must be confirmed by experienced Mitra Clip operators within the SEC. Subjects with primary MR must be at prohibitive surgical risk, while subjects with secondary MR must be symptomatic despite maximally-tolerated guideline-directed medical therapy and meet the Mitra Clip Indications for Use.

   Non-repairable cohort: Eligibility for this cohort is limited to subjects where the local site heart team deems the mitral valve anatomy is not suitable for TEER with Mitra Clip or does not meet Mitra Clip indications, which must be confirmed by experienced Mitra Clip operators from the SEC.

   Severe MAC cohort: Eligibility for this cohort is limited to subjects where the local site heart team deems the degree of MAC renders the subject unsuitable for mitral valve surgery.

   Severe MAC CAP cohort: Eligibility for this cohort is identical to the original Severe MAC cohort.
5. Age 18 years or older at time of consent.
6. Subject has been informed of the nature of the trial and agrees to its provisions, including the possibility of randomization to the Control group, complying with trial required testing, medications, and follow-up visits, and has provided written informed consent.

Exclusion Criteria:

1. Mitral valvular vegetation or mass.
2. Left Ventricle or Left Atrium thrombus.
3. Chest condition that prevents transapical access.
4. LVEF less than 25% assessed by the site based on a TTE obtained within 120 days prior to subject consent.

   Note: LVEF will be principally based on TTE and confirmed by the Echocardiography Core Laboratory.
5. LVEDD > 7.0 cm assessed by the site based on a TTE obtained within 120 days prior to subject consent.

   Note: A qualifying LVEDD must be confirmed by the Echocardiography Core Laboratory.
6. Prior surgical or interventional treatment of mitral valve involving implantation of prosthetic material (e.g. valve repair or replacement, or Mitra Clip).
7. Mitral pathoanatomy and LVOT anatomy deemed not suitable for Tendyne transcatheter mitral valve implantation.
8. Aortic valve disease requiring surgery or transcatheter intervention.
9. Tricuspid valve disease requiring surgery or transcatheter intervention.
10. Severe tricuspid regurgitation or severe right ventricular dysfunction.
11. Any surgical or interventional procedure within the period of 60 days prior to or planned procedure 60 days following subject registration.
12. Implant or revision of CRT device within 90 days prior to intended subject registration.
13. Myocardial infarction within 30 days prior to intended subject registration.
14. Symptomatic, unresolved multi-vessel or unprotected left main coronary artery disease (e.g., active ischemia) requiring stenting or CABG.
15. CVA within 6 months prior to intended subject registration.
16. Unresolved severe symptomatic carotid stenosis (> 70% by ultrasound).
17. Cardiogenic shock or hemodynamic instability requiring inotropes or mechanical support devices at the time of planned implant procedure.
18. Hypertrophic or restrictive cardiomyopathy, or constrictive pericarditis.
19. Any of the following: leukopenia, acute anemia, thrombocytopenia, history of bleeding diathesis, or coagulopathy if cannot be adequately treated.
20. History of endocarditis within 6 months of planned implant procedure.
21. Active systemic infection requiring antibiotic therapy.
22. Known hypersensitivity or contraindication to procedural or post-procedural medications (e.g., contrast solution, anti-coagulation or antiplatelet therapy) that cannot be adequately managed medically.
23. Subjects in whom TEE is contraindicated or high risk.
24. Known hypersensitivity to nickel or titanium.
25. Subject is undergoing hemodialysis due to chronic renal failure.
26. Subject has pulmonary arterial hypertension (fixed PAS >70mmHg). Note: If PAS > 70mmHg, site must provide documentation PAS is not fixed in order to be eligible.
27. Subject has COPD requiring continuous home oxygen therapy or chronic outpatient oral steroid use.
28. Subjects with non-cardiac comorbidities that are likely to result in a life expectancy of less than 12 months.
29. Modified Rankin Scale ≥ 4 disability.
30. Status 1 heart transplant or prior orthotopic heart transplantation.
31. Pregnant, lactating, or planning pregnancy during the clinical investigation follow-up period.

    Note: Female subjects of childbearing age should be instructed to use safe contraception (e.g. intrauterine devices, hormonal contraceptives: contraceptive pills, implants, transdermal patches hormonal vaginal devices, injections with prolonged release).
32. Currently participating in an investigational drug or another device trial that has not reached its primary endpoint.

    Note: Trials requiring extended follow-up for products that were investigational, but have since become commercially available, are not considered investigational trials.
33. Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements, or impact the scientific soundness of the clinical investigation results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2028-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Gorav Ailawadi, MD, Principal Investigator — University of Michigan; Jason Rogers, MD, Principal Investigator — University of California, Davis; Kyle Brunner, PhD, Study Director — Abbott Structural Heart; Paul Sorajja, MD, Principal Investigator — Allina Health System; Vinod Thourani, MD, Principal Investigator — Piedmont Healthcare and the Marcus Heart Valve Center
Locations (78):
- United States (73):
  - Princeton Baptist Medical Center, Birmingham, Alabama
  - UAB University Hospital, Birmingham, Alabama
  - Banner-University Medical Center, Phoenix, Arizona
  - HonorHealth Scottsdale Shea Medical Center, Scottsdale, Arizona
  - Baptist Health Medical Center, Little Rock, Arkansas
  - Fresno Heart Hospital, Fresno, California
  - University of Southern California University Hospital, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Sutter Medical Center, Sacramento, Sacramento, California
  - University of California - Davis Medical Center, Sacramento, California
  - San Diego Cardiac Center, San Diego, California
  - University of California at San Francisco, San Francisco, California
  - Stanford Health Care, Stanford, California
  - Los Robles Hospital and Medical Center, Thousand Oaks, California
  - University of Colorado Hospital, Aurora, Colorado
  - Manatee Memorial Hospital, Bradenton, Florida
  - Morton Plant Hospital, Clearwater, Florida
  - Delray Medical Center, Delray Beach, Florida
  - North Florida Regional Medical Center, Gainesville, Florida
  - Shands at the University of Florida, Gainesville, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Tallahassee Research Institute, Tallahassee, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Piedmont Heart Institute, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - St. Alphonsus Regional Medical Center, Boise, Idaho
  - Rush University Medical Center, Chicago, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Prairie Education & Research Cooperative, Springfield, Illinois
  - St. Vincent Hospital, Indianapolis, Indiana
  - Via Christi Regional Medical Center - St. Francis Campus, Wichita, Kansas
  - MedStar Health Research Institute, Balitmore, Maryland
  - University of Maryland Medical Center, Baltimore, Maryland
  - Adventist HealthCare White Oak Medical Center, Silver Spring, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - St. Luke's Hospital, Kansas City, Missouri
  - St. Louis University Hospital, St Louis, Missouri
  - The International Heart Institute of Montana, Missoula, Montana
  - Catholic Medical Center, Manchester, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Albany Medical College at Albany Medical Center, Albany, New York
  - South Shore University Hospital, Bay Shore, New York
  - Buffalo General Hospital, Buffalo, New York
  - New York Presbyterian Hospital/ Weill Cornell Medical Center, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Mission Health & Hospitals, Asheville, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Novant Health Heart and Vascular Research Institute, Charlotte, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Oklahoma Heart Institute at Utica, Tulsa, Oklahoma
  - Providence Heart & Vascular Institute, Portland, Oregon
  - Allegheny General Hospital - ASRI, Pittsburgh, Pennsylvania
  - UPMC Shadyside, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Baptist Memorial Hospital, Memphis, Tennessee
  - Centennial Medical Center, Nashville, Tennessee
  - St. Thomas Hospital, Nashville, Tennessee
  - Cardiothoracic & Vascular Surgeons, Austin, Texas
  - Baylor Scott & White Heart and Vascular Hospital, Dallas, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Memorial Hermann Hospital, Houston, Texas
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Swedish Medical Center - Heart & Vascular, Seattle, Washington
  - West Virginia University Hospital, Morgantown, West Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (5):
  - Ottawa Heart Institute, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Institut de Cardiologie de Montreal (Montreal Heart Institute), Montreal, Quebec
  - The Royal Victoria Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 103 subjects was registered in the Severe MAC cohort at a total of 37 sites with follow up through 12 months period
Period: Overall Study
Arm/Group | Severe Mitral Annular Calcification (MAC) Cohort
Started | 103
Completed | 73
Not Completed | 30
Not completed — Withdrawal by Subject | 2
Not completed — Missed visit | 5
Not completed — Death | 23

BASELINE CHARACTERISTICS:
Arm/Group | Severe Mitral Annular Calcification (MAC) Cohort
Number analyzed (Participants) | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 78 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57
  Male | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 99
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 101
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 3
  United States | 100
Hypertension [Count of Participants; unit: Participants] | 92

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Freedom From All-cause Mortality and Heart Failure Hospitalization (HFH)
Description: The primary endpoint for the Severe MAC cohort is freedom from all-cause mortality and heart failure hospitalization (HFH), evaluated against a performance goal of 43%.
Time Frame: 12 months post index procedure
Population: Attempted procedure (AP) population included subjects in whom a Tendyne procedure was attempted (initial incision for the Tendyne procedure)
Measure: Number (95% Confidence Interval); unit: percentage of participants -Kaplan Meier
Arm/Group | Severe Mitral Annular Calcification (MAC) Cohort
Number analyzed (Participants) | 103
percentage of participants -Kaplan Meier | 60.4 [50.2 to 69.2]
Statistical Analysis 1: Comparison: Severe Mitral Annular Calcification (MAC) Cohort; The null and alternative hypotheses are: H0: πD ≤ πPG H1: πD > πPG where πD is the true event rate for freedom from all-cause mortality and HFH at 12 months and πPG is the performance goal (PG); Test type: Other; p = 0.0002, one-sided 2.5% level of significance

2. Secondary Outcome: Percentage of Participants With Freedom From Mitral Regurgitation (MR) Severity > 1
Description: Freedom from MR > mild (1+) in severity at 1 month post index procedure among survivors.
  The null and alternative hypotheses are stated as:
  H0: PMR ≤ 1+ ≤ PPG H1: P MR ≤ 1+ > PPG where PMR ≤ 1+ is the proportion of subjects who have MR ≤ 1+ at 1 months post index procedure.
Time Frame: At 1 month post index procedure
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Severe Mitral Annular Calcification (MAC) Cohort
Number analyzed (Participants) | 98
percentage of participants | 100.0 [96.3 to 100.0]
Statistical Analysis 1: Comparison: Severe Mitral Annular Calcification (MAC) Cohort; The null and alternative hypotheses are stated as: H0: PMR ≤ 1+ ≤ PPG H1: P MR ≤ 1+ > PPG where PMR ≤ 1+ is the proportion of subjects who have MR ≤ 1+ at 30 days post index procedure; Test type: Other; p < 0.0001, Exact Binomial test; at a one-sided 2.5% level of significance

3. Secondary Outcome: Change in KCCQ Overall Score
Description: The Kansas City Cardiomyopathy Questionnaire (KCCQ) is a 23-item questionnaire developed to independently measure a patient's perception of their health status, which includes heart failure symptoms, impact on physical and social function, and how their heart failure impacts their quality of life. It includes questions on symptoms, physical limitations, social relationships, and emotional well-being. The KCCQ was administered by study personnel and completed by the subject. KCCQ scores range from 0-100, with 0 denoting the worst and 100 the best possible status. KCCQ-clinical summary score was average of domains- physical limitation and total symptoms (average of symptom frequency and symptom burden), and transformed to a single score which ranged from 0 (worst) -100 (the best possible status), where the higher score reflected better health status.
Time Frame: From Baseline at 12 Months
Population: Attempted procedure (AP) population included subjects in whom a Tendyne procedure was attempted (initial incision for the Tendyne procedure), were alive and with available data at 12 Months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Severe Mitral Annular Calcification (MAC) Cohort
Number analyzed (Participants) | 74
score on a scale | 69.9 (23.2)
Statistical Analysis 1: Comparison: Severe Mitral Annular Calcification (MAC) Cohort; The null and alternative hypotheses are: H0: D12M ≤ 0 H1: D12M > 0 Where D12M is the average change in KCCQ score from baseline at 12 months; Test type: Other; p < 0.0001, Paired t-test; at a one-sided 2.5% level of significance

4. Secondary Outcome: Change in Percentage of Participants With NYHA Class I & II
Description: New York Heart Association Classification (NYHA Class): NYHA class is an ordinal variable with higher classes indicating a worse degree of heart failure:
  Class I Patients with cardiac disease but without resulting limitations of physical activity.
  Class II Patients with cardiac disease resulting in slight limitation of physical activity. Patients are comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea, or anginal pain.
Time Frame: Change from Baseline at 12 Months
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Severe Mitral Annular Calcification (MAC) Cohort
Number analyzed (Participants) | 72
percentage of participants | 87.5 [77.6 to 94.1]
Statistical Analysis 1: Comparison: Severe Mitral Annular Calcification (MAC) Cohort; The null and alternative hypotheses are stated as: H0: PM12 = PB H1: PM12 ≠ PB where PM12 and PB represent the proportion of NYHA Classification I or II at 12 months and baseline, respectively; Test type: Other; p < 0.0001, McNemar; at a two-sided 5% level of significance

5. Secondary Outcome: Change in Six Minute Walk Test
Description: To evaluate the benefit of the Tendyne device, the distance walked at 12 months as measured by the 6MWT was compared with that from baseline. The six-minute walk test is a simple cardiopulmonary functional testing modality. Its straightforward nature allows for a non-specific, integrated assessment of the many systems involved during physical activity. Specifically, its results can assist in ascertaining the degree of functional impairment and potentially lead to modifications in therapy for some cardiovascular and pulmonary conditions.
Time Frame: From Baseline at 12 Months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Severe Mitral Annular Calcification (MAC) Cohort
Number analyzed (Participants) | 65
meters | 238.7 (109)
Statistical Analysis 1: Comparison: Severe Mitral Annular Calcification (MAC) Cohort; The null and alternative hypotheses are: H0: D12M ≤ 0 H1: D12M > 0 Where D12M is the average change in 6MWT distance from baseline at 12 months; Test type: Other; p = 0.0338, paired t-test; at a one-sided 2.5% significance level

ADVERSE EVENTS:
Time Frame: Through 1-year
Description: A detailed reporting of all deaths, adverse events and device deficiencies through 12 months in the Severe MAC cohort.
Arm/Group | Severe Mitral Annular Calcification (MAC) Cohort
All-Cause Mortality (participants affected / at risk) | 23/103
Serious Adverse Events (participants affected / at risk) | 81/103
Other Adverse Events (participants affected / at risk) | 3/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Severe Mitral Annular Calcification (MAC) Cohort (N=103)
Stroke or TIA (Nervous system disorders) | 4
Mitral Valve Reintervention (Surgical and medical procedures) | 5
Myocardial Infarction (Cardiac disorders) | 1
Bleeding (Injury, poisoning and procedural complications) | 39
Access Site and Vascular Complications (Vascular disorders) | 17
Cardiac Structural Complications due to Access Related Issues (MVARC) (Cardiac disorders) | 10
Acute Kidney Injury (MVARC) (Renal and urinary disorders) | 12
Respiratory Failure (>48 hour intubation) (Respiratory, thoracic and mediastinal disorders) | 9
Arrhythmia or Conduction Disturbance (Cardiac disorders) | 41
Endocarditis (Infections and infestations) | 4
Device Thrombosis (Vascular disorders) | 3
Emergency Surgery or Intervention during Index Procedure (Surgical and medical procedures) | 5
Other (General disorders) | 51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Severe Mitral Annular Calcification (MAC) Cohort (N=103)
PERICARDITIS (Cardiac disorders) | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 1
HYPOTENSION (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-05-05): https://cdn.clinicaltrials.gov/large-docs/74/NCT03433274/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-20): https://cdn.clinicaltrials.gov/large-docs/74/NCT03433274/SAP_001.pdf